CLINICAL TRIAL: NCT00061646
Title: A Phase II Single-Arm Study Evaluating the Safety and Effectiveness of ABT-510 Plus Combination Chemotherapy in Subjects With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Effectiveness of ABT-510 Plus Combination Chemotherapy in Subjects With Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment suspended based upon interim analysis; subjects allowed to stay on study until disease progression.
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-429
Record Dates: First submitted 2003-06-02; First posted 2003-06-04 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Stage IIIb with pleural effusion or IV NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-510/Thrombospondin-1 mimetic
Drug: Carboplatin/Taxol

SUMMARY:
The primary objective of this Phase II study is to assess the safety, pharmacokinetics and effectiveness of ABT-510 in combination with standard carboplatin/paclitaxel chemotherapy in subjects with stage IIIb or IV NSCLC.

ELIGIBILITY:
Inclusion Criteria

* The subject is at least 18 years of age.
* The subject has histologically or cytology documented Stage IIIB with pleural effusion or Stage IV NSCLC. The subject must have measurable disease (RECIST Criteria for Tumor Response).
* The subject has not received first line therapy for treatment of NSCLC.
* The subject must not be pregnant or lactating and all subjects (male and female) must use a contraceptive method deemed acceptable by the investigator while in the study and for up to two months following completion of therapy.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
* The subject is able to self-administer or has a caregiver who can reliably administer SC injections.
* The subject must have adequate bone marrow, renal and hepatic function as follows:

  * Bone marrow: White blood cell count (WBC) >= 3,000/mm3; Platelets; >= 100,000/mm3; Hemoglobin >= 9.0 g/dL;
  * Renal function: Serum creatinine <= 2.0 mg/dL;
  * Hepatic function: Bilirubin <= 1.5 mg/dL; AST and ALT <= 1.5 X the upper normal limit (ULN); unless liver metastases are present, then AST and ALT <= 5.0 x ULN.
* The subject has voluntarily signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved consent prior to any study specific procedures.

Exclusion Criteria

* The subject has a history of or currently exhibits Central Nervous System (CNS) metastasis. Brain MRI within 28 days of enrollment is required to confirm absence of CNS metastases.
* The subject is receiving therapeutic anticoagulation therapy. Low dose anticoagulation for catheter prophylaxis will be permitted; PT/PTT must be within normal limits.
* The subject has a history of or currently exhibits clinically significant cancer related events of bleeding (e.g., hemoptysis). The subject has a recent history of (within 4 weeks from Study Day 1) or currently exhibits other clinically significant events of bleeding.
* The subject has received investigational therapy within four weeks prior to study drug administration.
* The subject exhibits evidence of clinically significant uncontrolled condition(s) and/or is considered by the investigator to be unable to tolerate the proposed treatment or procedures.
* The subject has previous or current malignancies at other sites, with the exception of: Adequately treated in situ carcinoma of the cervix uteri; Basal or squamous cell carcinoma of the skin; Previous nonpulmonary malignancy confined and surgically resected with no evidence of active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-03

PRIMARY OUTCOMES:
Progression free survival | One year

SECONDARY OUTCOMES:
Overall survival | One year
Response rate | One year

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott
Locations (4):
- United States (4):
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - The West Cancer Clinic, Memphis, Tennessee
  - University of Wisconsin, Madison, Wisconsin